CLINICAL TRIAL: NCT06801314
Title: Effect of Early Mobilization Exercises Guided by Wearable Technology on Functional Capacity After Coronary Artery Bypass Graft
Brief Title: Effect of Early Mobilization Exercises After Coronary Artery Bypass Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Ali Mohamed Awad Allah, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005234
Record Dates: First submitted 2025-01-16; First posted 2025-01-30 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Bypass Graft CABG
Keywords: CABG
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: patients will be randomly assigned into three groups, group A will receive usual care , group B will receive usual care in addition to aerobic exercise and group C will receive usual care in addition to resisted exercise
Who Masked: Participant, Investigator
Masking Description: double blinded(participant ,, investigator )
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (A) usual care (Active Comparator): patients in this group will receive usual care including moibilizations and breathing exercise
- study group (B)aerobic exercise (using cycle ergometer) in addition to usual care (Experimental): Patients in this group will be received usual care and cycle ergometer aerobic exercise
  Interventions: Other: aerobic exercise using cycle ergometer in addition to usual care
- study group(C)resisted exercise group (using weights and dumbbells) in addition to usual care (Experimental): Patients in this group will be received usual care and resisted exercise
  Interventions: Other: resisted exercise using weights and dumbbells in addition to usual care

INTERVENTIONS:
Other: aerobic exercise using cycle ergometer in addition to usual care — aerobic exercise group):Patients in this group will be received usual care and cycle ergometer aerobic exercise Mood of exercise: continuous aerobic exercise
  * Modality of exercise: cycle ergometer
  * Intensity of exercise: low to moderate intensity and HR (calculated as recommended by the American College of Sports Medicine (ACSM) and tolerated up to 20-30 bpm above the resting HR), BP, SpO2 and rate of perceived exertion through the Borg Scale (10-13) will be monitor during cycling
  * Duration: 15-20 min including 5 min warm up and 5 min cool down and working phase from 5-10 min
  * Frequency: daily until discharge aerobic exercise group guided by wearable artificial intelligence ECG monitor to real-time support, guide and stop exercise when there is any adverse events will occur.
  Arms: study group (B)aerobic exercise (using cycle ergometer) in addition to usual care
Other: resisted exercise using weights and dumbbells in addition to usual care — resisted exercise group): Patients in this group will be received usual care and resisted exercise
  * Mode: resisted exercise
  * Modality: dumbbells or sand bags tied around main groups of muscles for upper and lower limbs Intensity of exercise: the load that the patient can lift for 10-12 repetition at RPE of 10-13 and 1-2 sets resisted exercise group guided by wearable artificial intelligence ECG monitor to real-time support, guided and stop exercise when there is any adverse events will occur.
  Arms: study group(C)resisted exercise group (using weights and dumbbells) in addition to usual care
Other: usual care using mobilization and breathing exercise — mobilization and breathing exercise

SUMMARY:
purpose: This study aims to assess the effects of early mobilization exercises guided by wearable technology on functional capacity after coronary artery bypass graft Methods: Patients will be randomly assigned into three groups: Group A will receive usual care, Group B will receive usual care in addition to aerobic exercise, and Group C will receive usual care in addition to resistance exercise. both the aerobic exercise group and the resistance exercise group will be guided by wearable artificial intelligence ECG monitors for real-time support and guidance, and they will stop exercise when any adverse events occur.

Exercises will be started early from post operative CABG until patients discharge and measurements will be taken at baseline and before discharge

DETAILED DESCRIPTION:
A) Procedure for evaluation and training

Equipment:

The following instruments will be used:

* Pulse oximeter: It will be used for measuring oxygen saturation and Heart rate before, during, and after sessions and during exercise test
* Intelligent cardiac monitor: used during 6MWT to detect any adverse events during and immediately after the test and also be used during sessions
* Rating of perceived exertion: to estimate effort and exertion during the test and working phase.
* Cycle ergometer: upper and lower pedaling machine will be adjusted to suit all patients' height during exercise sessions
* Dumbbells and weights will be used during exercise sessions Exercise (treatment) procedures
* Group (A): (usual care group):

Start early mobilization exercises and deep breathing exercises with wound support daily

* Group (B): (aerobic exercise group): Patients in this group will receive usual care and cycle ergometer aerobic exercise Mood of exercise: continuous aerobic exercise
* Modality of exercise: cycle ergometer with upper and lower pedaling at the same time with adducted shoulders.
* Intensity of exercise: low to moderate intensity and HR (calculated as recommended by the American College of Sports Medicine (ACSM) and tolerated up to 20-30 bpm above the resting HR), BP, SpO2 and low to moderate rate of perceived exertion through the Borg Scale (10-13) will be monitored during cycling
* Duration: 15-20 min, including 5 min warm-up, 5 min cool down and a working phase from 5-10 min
* Frequency: Daily until discharge
* Group (C): (resisted exercise group):

Patients in this group will receive usual care and resisted exercise

* Mode: Resisted exercise
* Modality: dumbbells or sandbags tied around main groups of muscles Resistance exercises consisted of muscle training with dumbbells for the upper limb (UL) (biceps, triceps, and shoulder flexors) and sandbags for the lower limb (LL) (quadriceps, hamstrings, abductors, and calves).

Intensity of exercise: the load that the patient can lift for 10-12 repetitions at RPE of 10-13 and 1-2 sets Both the aerobic exercise group and the resistance exercise group will be guided by wearable artificial intelligence ECG monitors to provide real-time support and guidance and stop exercise when adverse events occur.

ELIGIBILITY:
Inclusion Criteria:

1-post -operative clinically stable patients with hemodynamic stability through measurement of respiratory rate( >8<30) breaths/min , Heart rate (>40<130) beats /min , Spo2>90% 2-both lower limbs will be physically functional 3-CABG surgery 4-Their age will be ranged from 45-65 years old

- Exclusion Criteria:

1. Respiratory insufficiency after surgery manifesting hypoxemia with partial pressure of oxygen in arterial blood <60 mmHg
2. Cardiogenic shock
3. acute renal failure
4. contra-indicated to submaximal exercise test
5. cardiac arrhythmia
6. locomotor/neurological limitation to ambulation
7. physiological compensatory tachycardia in case of (anemia, high tempreture and infection)
8. high blood pressure at rest (systolic blood pressure >160mmHg or diastolic blood pressure >100 mmHg -

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Functional capacity | at baseline before intervention and 1 week after intervention
  Functional capacity: It will be assessed by 6MWT test. According to the American Thoracic Society,

SECONDARY OUTCOMES:
Heart rate variability | at baseline before intervention and 1 week after intervention
  Assessed by AI- ECG cardiac monitor to detect variation in time between subsequent heart beats(R-R interval) at base line and before discharge
- Muscle strength | at baseline before intervention and 1 week after intervention
  It will be assessed by chair stand test by patient standing /sitting with arms crossed at the wrists against the chest, the numbers of stands in 30s is recorded
- Kinesiophobia | at baseline before intervention and 1 week after intervention
  It will be assessed by Tampa Scale 11 (TSK-11) 11-item, 2-factor structure best fit the data. The first factor, somatic focus, consisted of 5 items, while the second factor, activity avoidance, was comprised of 6 items
- Functional independence | at baseline before intervention and 1 week after intervention
  It will be assessed by Barthel index score to ascertain the patients' abilities to perform activities of daily living
- Length of hospital stay | after 1 week of intervention
  is a promising alternative for costs management and efficient consumption of hospital recourses
- Adherence | after 1 week of intervention
  Adherence to the intervention was defined as completing at least 75% of the exercises and consultations
- Patient Safety | after 1 week of intervention
  Patient safety ( the exercise session will be terminated if any adverse events or arrhythmia occur in patients, which leads to a change in ECG waves in the mobile screen ) eg: Atrial fibrillation causes the absence of the p-wave and a narrow QRS complex.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Mahdy Ahmad, A.professor, Study Director — Cairo University; NESREEN G EL_NAHAS, professor, Study Chair — Cairo University; Sara Ali AWAD ALLAH, Assistant professor, Principal Investigator — Cairo University; Alaa Eldin Abdelaty Bahy, consultant, Study Director — Cairo University
Locations (1):
- Faculty of physical therapy, Cairo university, Giza, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No